CLINICAL TRIAL: NCT01702935
Title: Oogonial Stem Cell Isolation in Ovarian Insufficiency Patients
Brief Title: Ovarian Stem Cells From Women With Ovarian Insufficiency
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120212; 12-CH-0212
Record Dates: First submitted 2012-10-06; First posted 2012-10-10 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2017-09-21

CONDITIONS: Infertility
Keywords: Ovarian Failure; Premature Ovarian Failure; Infertility; Primary Ovarian Insufficiency; Stem Cells
MeSH Terms: conditions — Infertility; Primary Ovarian Insufficiency

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Primary ovarian insufficiency (POI) is a condition that affects ovary function. It means that the ovaries are not able to function at a level appropriate for a woman's age. Previously, it was thought that women had only a fixed number of eggs that were lost each month until none were left at menopause. However, recently, stem cells have been found in the ovaries of adult women. These stem cells may be able to make new eggs. Studying these cells may help women with POI in the future. Researchers want to collect ovarian tissue from women with POI to investigate ovarian stem cells.

Objectives:

- To collect ovarian tissue from women with primary ovarian insufficiency.

Eligibility:

- Women between 18 and 50 years of age with primary ovarian insufficiency.

Design:

* Participants will be screened with a physical exam and medical history. They will also have a full gynecological exam. They will provide blood and urine samples.
* Participants will donate ovarian tissue for study. It will be collected through outpatient surgery. The surgery will take either half of an ovary or a full ovary.
* Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
Early loss of human ovarian function results in a clinical condition known as primary ovarian insufficiency (POI) or premature ovarian failure (POF). This devastating condition renders women unable to have their own genetic child in more than 95% of cases (1), as well as failure of hormonal production by the ovary that is critical in maintaining bone health, restful sleep, and quality of life. Indeed, in more carefully designed studies where control groups were used, only 1.5% of POI patients became pregnant (2-8), which may more accurately represent the true fertility rate in this population. Currently, fertility treatments for these patients are primarily to use an egg donated from a young woman

Until recently, it was thought that women were born with a limited number of eggs, which were slowly depleted each month until exhaustion at the time of menopause. However, recent studies have suggested that new eggs can be made from adult stem cells in the ovary. (1, 2) These ovarian stem cells could be transplanted into a recipient mouse, who then delivered donor derived offspring (3). Recently, ovarian germline stem cell (i.e., oogonial stem cell) isolation has been reported from human ovaries (12).(4). However, it is not known if oogonial stem cell problems play a part in diseases such as premature ovarian failure or diminished ovarian reserve.

The goal of this protocol is to characterize oogonial stem cells in patients with primary ovarian insufficiency (POI)/failure (POF) and diminished ovarian reserve (DOR). There will be three groups in this study: patients with POI or POF undergoing ovarian biopsy by laparoscopy, patients with POI or POF undergoing clinically indicated abdominal surgery that provides access to the ovaries, and patients over 18 undergoing clinically indicated ovarian surgery (with or without POI or POF). Ovarian biopsies will be harvested by laparoscopy or at the time of indicated surgery, and oogonial stem cells will be isolated in the laboratory and characterized.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subject is able to give consent/assent to participate in the protocol.

Listed below are acceptable medical conditions for inclusion in this protocol:

* Females older than 18 years with POI, POF, or DOR, undergoing ovarian biopsy by laparoscopy or clinically indicated abdominal surgery that provides access to the ovaries

  * Clinical etiologies of POI may include, but are not limited to, idiopathic, autoimmune, chemotherapy related, or Turner s syndrome
  * Subjects must have a diagnosis of premature ovarian failure or diminished ovarian reserve as defined by both:

    1. Early follicular phase FSH >15 IU/L
    2. AMH <0.16 ng/ml or below the level of detection for the assay used
* Females older than 18 years, with or without POI or POF, undergoing clinically indicated ovarian surgery

EXCLUSION CRITERIA:

Unable to comprehend the investigational nature of the protocol participation

Positive pregnancy test

Anticoagulation or known coagulopathy

Ovarian cancer

History of a previous laparoscopy or laparotomy revealing abdominal adhesions that would preclude ovarian biopsy

Previous bowel surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-09-19; Study Completion 2017-09-21

PRIMARY OUTCOMES:
The immediate aim of this protocol is to characterize oogonial stem cells in patients with primary ovarian insufficiency and diminished ovarian reserve.

CONTACTS AND LOCATIONS:
Overall Officials: Alan H DeCherney, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] van Kasteren YM, Schoemaker J. Premature ovarian failure: a systematic review on therapeutic interventions to restore ovarian function and achieve pregnancy. Hum Reprod Update. 1999 Sep-Oct;5(5):483-92. doi: 10.1093/humupd/5.5.483. PMID 10582785
- [Background] Anasti JN, Kimzey LM, Defensor RA, White B, Nelson LM. A controlled study of danazol for the treatment of karyotypically normal spontaneous premature ovarian failure. Fertil Steril. 1994 Oct;62(4):726-30. doi: 10.1016/s0015-0282(16)56996-9. PMID 7926080
- [Background] Nelson LM, Kimzey LM, White BJ, Merriam GR. Gonadotropin suppression for the treatment of karyotypically normal spontaneous premature ovarian failure: a controlled trial. Fertil Steril. 1992 Jan;57(1):50-5. doi: 10.1016/s0015-0282(16)54775-x. PMID 1730330